CLINICAL TRIAL: NCT04290117
Title: Chronobiological and Acceptance and Commitment Based Training for the Successful Handling of Stress in the Workplace. A Randomised Crossover Clinical Study
Brief Title: Chronobiological and ACT-based Training to Handle Stress at Work
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Principal Investigator, Carolin Reichert, Principal Investigator, Psychiatric Hospital of the University of Basel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01318
Record Dates: First submitted 2019-09-05; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Stress
Keywords: Sleep Hygiene; Morning Light; Acceptance and Commitment Training
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ACT-Chrono (Experimental): First Acceptance and Commitment (ACT) training, followed by chronobiological training
  Interventions: Behavioral: Acceptance and Commitment Training; Behavioral: Sleep Hygiene and bright light in the morning
- Chrono-ACT (Experimental): First chronobiological training, followed by ACT training
  Interventions: Behavioral: Acceptance and Commitment Training; Behavioral: Sleep Hygiene and bright light in the morning
- Chrono (Other): First no training, followed by chronobiological training
  Interventions: Behavioral: Sleep Hygiene and bright light in the morning
- ACT (Other): First no training, followed by ACT training
  Interventions: Behavioral: Acceptance and Commitment Training

INTERVENTIONS:
Behavioral: Acceptance and Commitment Training — During the ACT-based intervention, participants will get 4 training sessions in groups, once a week for an hour. Additionally, participants will be asked to implement behavioural exercises such as mindfulness and value-based exercises into their daily schedule.
  Arms: ACT; ACT-Chrono; Chrono-ACT
Behavioral: Sleep Hygiene and bright light in the morning — During the chronobiological intervention, participants will get 4 training sessions in groups, one hour per week. Additionally, they will use a daylight lamp at home, for 30 minutes per day after waking up.
  Arms: ACT-Chrono; Chrono; Chrono-ACT

SUMMARY:
The aim of the present project is to combine "Acceptance and Commitment Therapy" and "sleep hygiene + light-therapy (so-called chronotherapy)" serially in a sample of employees to reduce levels of subjective exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* working in an office mainly (i.e., > 60% of work time)
* Age: ≥18 years old
* Sex: male and female individuals
* Ownership of cell phone with internet connection
* informed consent as documented by signature

Exclusion Criteria:

* diseases of the retina or related diseases such as diabetes mellitus
* taking drugs which heighten photosensitivity
* inability to understand and follow procedures in German

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in subjective exhaustion measured by the German Version of the Shirom-Melamed Burnout Measure | approx. every two weeks, and at follow up (i.e., approx. 5 weeks after last training session)
  Overall mean score as well as three subscales of Shirom-Melamed Burnout Measure ( P = physical fatigue; E= emotional exhaustion; and C= cognitive weariness, each ranging from 1-7).
  Note: Higher scores indicate higher levels of exhaustion (overall as well as on each scale P, E and C)

SECONDARY OUTCOMES:
Change in Subjective well-being as assessed by General Health Questionnaire (GHQ-12) | approx. every two weeks, and at follow up (i.e., approx. 5 weeks after last training session)
  Sum over twelve items, higher scores indicate worse psychological well-being
Change in subjective well-being as assessed by the Patient Health Questionnaire (PHQ-D) | approx. every 4 weeks
  Sum over each of the subscales assessing somatic, depressive, anxiety and stress symptoms. The subscale assessing panic symptoms, alcohol abuse and intake of medication will be categorically evaluated.
Change in quality of circadian rhythm | Actimetric devices are worn during 2 x 28 days continuously. The outcome of actimetric data are aggregated per person and training episode
  Actimetric devices are worn during 2 x 28 days continuously. These devices store the amount of activity in a resolution of 30 Hz 24/7. For data analyses, these activity data will be aggregated to three values (stability, variability and relative amplitude) per participant and training episode by non-parametric circadian rhythm analyses; higher values indicate higher stability, variability and amplitude
Change in subjective and objective sleep quality: Pittsburgh Sleep Quality Index (PSQI) | PSQI is collected approx. every four weeks and at follow up (i.e. approx 5 weeks after last training), the single question and actimetric data are measured daily
  Subjectively assessed by the Pittsburgh Sleep Quality Index (PSQI, higher scores indicate worse subjective sleep quality), by a single question about sleep quality (higher scores indicate worse quality) and by actimetric analyses
Change in Subjective sleepiness in the morning | KSS is measured daily
  Measured by Karolinska Sleepiness Scale (KSS), higher scores indicate higher sleepiness
Change in daytime subjective sleepiness | ESS approx every four weeks
  Measured by Epworth Sleepiness Scale (ESS): higher scores indicate higher sleepiness
Change in Chronotype | approx. every 4 weeks and at follow up (i.e., approx. 5 weeks after last training session)
  Measured by a short version of the Munich Chronotype Questionnaire, higher scores indicate a later chronotype
Change in Burnout severity | every 4 weeks
  Measured by Maslach Burnout Inventory using sumscores of the subscales emotional exhaustion, depersonalization and personal achievement. Higher scores indicate higher exhaustion, depersonalization and better personal achievement
Change in Absences | Assessed daily
  Numbers of days absent if available from the employer
Change in Implementation of treatment | approx. every two weeks, and at follow up (i.e., approx. 5 weeks after last training session)
  Questions about frequency implementation of treatment in daily life

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Reichert, PhD, Principal Investigator — Centre for Chronobiology
Locations (1):
- Centre for Chronobiology, UPK Basel, Basel, Switzerland